# 知情同意书

项目名称: 髌腱联合筋膜手法协调中心点的体外冲击波治疗髌腱炎的临床疗效: 一项随机对照试验

研究单位:中山大学孙逸仙纪念医院

本中心主要研究者: 柯松坚

尊敬的研究参与者:

我们邀请您参加一项研究,项目名称是"髌腱联合筋膜手法协调中心点的体外冲击波治疗 髌腱炎的临床疗效:一项随机对照试验"。

本知情同意书将详细讲述这项研究的相关信息、目的、研究流程、任何潜在的获益和风险 以及您的权利等内容,在您做出参加这项研究的决定之前,请您仔细阅读以下信息,如果有任 何疑问请向研究医生或研究人员提出。您可以与家人以及朋友讨论,并有充足的时间来考虑。 如果您正在参加别的研究,请告知您的研究医生或研究人员。

如果您已经详细了解了这项研究,并决定参加,您需要签署这份知情同意书,我们将提供您一份已签署的知情同意书副本。

#### 一、为什么进行这项研究?

1、研究背景:

髌腱炎常见髌骨下极(髌腱近端)疼痛,严重时可牵涉至髌下区域;同时可伴随肿胀、膝关节无力等症状。临床上髌腱炎的保守治疗手段包括服用抗炎药、局部注射、支具固定、运动疗法、手法治疗、肌内贴扎技术、体外冲击波疗法(ESWT)、激光和超声波治疗等,但目前证据显示口服非甾体药物的治疗效果维持较短,而离子电渗疗法、按摩、电疗、运动锻炼和皮质类固醇注射等治疗有较长期效果但容易复发。这些治疗手段中大部分都是针对髌腱区域组织进行消炎止痛的,只有体外冲击波针对髌腱去进行刺激性治疗,刺激肌腱的修复和组织再生。

近年来,体外冲击波疗法(ESWT)以其修复作用在治疗髌腱炎等肌腱病中的应用激增。冲击波疗法被认为可以通过新生血管形成、细胞增殖和抗炎作用等多种机制刺激慢性肌腱病的组织修复和再生,并减轻局部的疼痛和降低敏感性。国内外大部分研究通过对髌腱周围痛点进行治疗,可有效缓解疼痛和提高膝关节功能,是治疗髌腱炎的有效手段,但

部分长期疗效尚未明确。意大利筋膜手法(fascial manipulation, FM)基于身体一体化理论,从筋膜相互影响的原则,采用结构化的评估以识别髌腱周围特定筋膜致密化区域,消除筋膜致密化,恢复筋膜组织生理张力并促进层间正常滑动,在减轻髌腱炎患者患膝负荷、改善患侧下肢生物力学、防止疼痛加重方面体现出非常大的潜力。 因此,筋膜手法也被证实可缓解髌腱炎疼痛。

体外冲击波治疗(ESWT)治疗原理是导子通过对靶区的高速震动进行松解筋膜,可同样改善筋膜链的异常张力。因此本研究探讨基于筋膜理论,采用髌腱联合筋膜手法协调中心点进行体外冲击波治疗,观察其治疗效果是否优于单纯髌腱痛点治疗方案,通过改变筋膜异常张力以维持更长时间的治疗效果。

#### 2、研究目的:

评估髌腱联合筋膜手法协调中心点体外冲击波治疗髌腱炎在缓解疼痛、改善膝关节功能障碍方面的有效性和持久性,明确在髌腱炎的冲击波治疗中联合协调中心点的治疗思路是否优于传统的痛点(单纯髌腱)治疗,探究髌腱炎冲击波治疗中的一种更加持久高效的方法。

**3**、本研究已获得中山大学孙逸仙纪念医院医学伦理委员会的批准,伦理委员会是一个保护研究参与者权益的组织。

#### 二、研究项目介绍

- 1、研究设计:本研究为单中心研究,计划在本中心纳入 38 名研究参与者。研究起止时间为 2025 年 10 月至 2026 年 12 月。
  - 2、参加本研究需要符合的条件:
  - 1) 您必须符合下列所有标准才能入选:
  - A. 年龄为 18 至 45 岁的成年人;
  - B. 符合《实用运动医学》(2023版) 髌腱炎诊断标准;
  - C. 膝关节疼痛 VAS 评分≥3 分及≤7 分;
  - D. 无其他影响下肢力量或行走的骨科或神经系统疾病;
  - E. 自愿签署知情同意书,并能够配合本研究的治疗和随访。
  - 2) 如果您符合下列条件之一,将不能参加本研究:
  - A. 一年内膝关节手术史;
  - B. 存在其他原因导致的膝关节前侧疼痛,或有累及膝关节疼痛性疾病或影响关节的疾病(包括但不限于:一过性滑膜炎、骨结核、骨肿瘤、急性创伤性关节炎、化脓性关节炎、类风湿性关节炎、代谢性骨病、银屑性关节炎、痛风性关节炎、骨坏死、强直性脊柱炎或

活动性感染等);

- C. 存在因其他原因引起的膝关节的慢性疼痛(如带状疱疹后神经痛、骨质疏松等):
- D. 使用冲击波治疗的禁忌症,例如:下肢深静脉血栓、出血性疾病或凝血功能障碍、妊娠、认知功能障碍等:
- E. 有癌性肿瘤、严重支气管扩张、急性化脓性炎症、高烧、活动性肺结核、心力衰竭、 严重贫血、脑血管疾病,或体内植入心脏起搏器等
- F. 由于其他健康问题无法参与试验,如突发严重外伤、突发严重传染性疾病等。

#### 三、这项研究是怎样进行的?

- 1、签署知情同意书
- 2、进行研究的入组筛选,研究医生将收集您的现病史、既往史、体格检查、患侧膝关节的 VAS 评分(疼痛情况)、Lysholm 膝关节评分(功能情况)和超声下评估髌腱厚度。
- 3、研究分组及治疗。本研究为随机对照双盲设计,双盲是指您和研究人员均不清楚您的分组和接受的研究干预。

如您满足入选条件,您将按 1:1 的比例随机编入试验组或对照组,按照研究方案接受相应的治疗。

试验组:

第1天行第一次髌腱联合筋膜手法协调中心点体外冲击波治疗,1周后行第二次髌腱联合筋膜手法协调中心点体外冲击波治疗,2周后行第三次髌腱联合筋膜手法协调中心点体外冲击波治疗。

对照组:

第1天行第一次单纯髌腱体外冲击波治疗,1周后行第二次单纯髌腱体外冲击波治疗,2周后行第三次单纯髌腱体外冲击波治疗。

#### 4、 访视随访

您需在全部治疗完成后 1 个月和 3 个月时完成随访, 医生将在全部治疗完成后 1 个月和 3 个月时对您进行电话随访。按照方案要求, 您的医生将安排您进行如下随访检查项目:

访视 1,全部治疗完成后 1 个月

- 病史、体格检查
- VAS 评分
- Lysholm 膝关节评分

访视 2,全部治疗完成后 3 个月

- 病史、体格检查
- VAS 评分
- Lysholm 膝关节评分
- 5、 需您配合的事项

研究期间,您需向研究医生如实告知您的病情,以及您目前正在使用的其他治疗药物,如果您的身体和精神方面出现不适反应,请您及时告知医生,无论这种改变是否与研究有关。请您务必告知您的医生您目前正在使用以及在研究期间使用的任何其他药物。如需其他治疗,请事先与您的医生联系,以获得正规医学指导。

#### 四、可选择的其他替代治疗

参加本研究是完全自愿的,如果您不参加、或在研究的任何阶段选择退出,您可以选择接受替代治疗。替代治疗方法包括:口服抗炎药、局部注射、支具固定、运动疗法、手法治疗、肌内贴扎技术、激光和超声波治疗等。您可以和您的医生在决定是否参加本研究前讨论具体的替代治疗方法。

# 五、与本研究相关的费用情况

● 本研究中所使用的膝关节 VAS 评分和 Lysholm 膝关节评分、髌腱的超声厚度评估等检查费用免费。冲击波治疗为临床指南推荐的疗法,为常规治疗项目,费用需要您自行承担。参加本研究不会额外增加您的经济负担。

#### 六、您的预期受益

参与本研究,您的疾病有可能得到缓解,但也有可能达不到预期的效果,甚至出现疾病进展;所接受的治疗和检查也许不能使您直接受益,但您的参与有助于医学对此类疾病的进一步研究和认识,有希望在未来提高疾病的诊疗水平。

## 七、可能给您带来的不便、不适和风险

本研究干预有可能给您带来不适或者出现不可预知的甚至是严重的不良反应。根据现有的研究数据,使用冲击波治疗可能会出现以下不良反应:

- 1. 治疗后治疗区域皮肤破损、红肿或瘀斑;
- 2. 治疗过程中患者出现痛性晕厥;
- 3. 治疗后治疗区域出现神经刺激感和皮肤瘙痒;
- 4.治疗后短期内疼痛加重。

本研究需要您配合回院随访,可能会占用您一定的时间。

研究过程中可能问及一些敏感类问题,如果您觉得有不适的话题,可以拒绝回答。

因此,如果研究过程中您出现任何不适,请及时告知您的医生,医生会给您提供及时的诊断及必要的医疗和建议。

#### 妊娠风险

由于不知道冲击波治疗对胎儿的影响,您在加入研究的时候不能是孕期,且您在研究过程中也不得怀孕,这非常重要。如果您已怀孕、准备怀孕,则您不得参与本研究。

如果您是女性研究参与者,具有生育能力,在您开始研究之前,您需要先进行妊娠测试。

如果您是女性受试者,具有生育能力,请您在研究期间使用可靠的避孕方法进行避孕。研究医生会告诉您哪些是可接受的避孕方法。建议采用下列避孕方法:带有或不带有杀精剂(杀死精子的药物)的避孕套、带有杀精剂的阴道隔膜或宫颈帽,或宫内节育装置(安装在女性子宫内的避孕小装置)。在无保护性性行为发生后采取的紧急避孕措施,如紧急避孕药,不能作为常规避孕方法运用。如果您在参与研究期间发现妊娠测试结果呈阳性,您应立即告知研究医生。如果确认您怀孕,您需要立即停止冲击波治疗,并按方案要求接受进一步随访和检查,研究医生可能会要求您退出研究。研究医生可能会在研究期间收集关于您的妊娠相关信息。

## 八、研究相关损害的处理和赔偿

如果发生研究相关的损害,研究者会进行积极的治疗,本中心将依法承担相关的医疗费用 及补偿费用。本研究未购买临床试验保险。

#### 九、保密的措施

本研究的结果只用于科研目的,因此您参加研究及研究中您的个人资料均属保密,将依照 法律规定得到保护,不会泄露您的名字和身份,您的姓名不会出现在任何研究报告和公开出版 物中。政府管理部门、医院伦理委员会、研究者等如因工作需要,按规定有权接触您所有的研 究资料,包括临床观察表、研究数据等。

## 十、研究终止

参加研究期间,您可以随时退出研究而不需要理由,您的决定不会对您继续接受医学治疗 产生任何影响。您的医生也可能由于下列原因停止您继续参加研究:

- 您没有遵循研究医生的指导和要求;
- 疾病进展或出现不可耐受的不良反应,研究医生认为继续参加研究会对您造成危害;
- 您接受了本项研究不允许的治疗;
- 研究医生、伦理委员会或政府管理部门要求停止本项研究。

当您退出研究或研究终止时,研究医生将与您讨论后续的诊疗措施。

# 十一、您的权利

本研究已获得中山大学孙逸仙纪念医院医学伦理委员会的审核、同意,方案设计合乎伦理要求,这将会保证您的权益在本研究中不受侵犯。

您参加本研究完全是自愿的,您可以拒绝参加或在任何时间退出,而不会遭到歧视或报复,您的医疗待遇与权益也不会受影响。如果您退出研究,为了安全考虑,您在退出时应该完成一些相应的医学检查。如果研究期间医生认为您不适合继续参加时,为保护您的利益,医生有权决定中止您继续参加本研究。另外,研究期间,您可以随时了解与研究有关的信息资料。如果我们获知了一些关于本研究的最新信息也将及时通知您,让您决定是否继续参加研究。

在研究期间,一旦出现任何不适或病情加重,请立即通知您的研究医生,我们会及时采取相应的医疗措施。对于发生的与研究相关的不良事件,研究者会进行积极的治疗。

## 十二、详细联系信息

如果关于参加本研究您有任何担忧或疑问,或如果您在参加本研究时经历任何异常反应, 或如果发生紧急情况,您可以直接与研究者联系:

研究人员: 柯松坚 联系电话: (020) 81332732 手机号码: 13760623229

如果您有与自身权利/权益相关的任何问题,或者您想反映治疗过程中遭遇的困难、不满和忧虑,或者想提供有关的意见和建议,请联系中山大学孙逸仙纪念医院医学伦理委员会,联系电话: 020-81332587,电子邮箱: sysyx11wyh@163.com。

# 知情同意书•同意签字页

# 研究参与者声明

我本人已认真阅读该知情同意书,研究人员已向我做了详尽说明并解答了我的相关问题, 我已充分知晓了以下内容:

- (1) 作为研究参与者,我将遵守研究参与者须知要求,自愿参加本研究,并与研究人员充分 合作,如实、客观地向研究人员提供参加本研究前的健康状况及相关情况。
- (2) 我同意中山大学孙逸仙纪念医院基于科学研究的目的查阅我的医学资料和研究结果。我 了解本研究的结果只用于科研目的,除外政府管理部门、伦理委员会、研究者等,我参 加研究及研究中的个人资料均属保密,将依照法律规定得到保护。
- (3) 我自愿参加本研究,如果在研究中出现与研究相关的不良反应,我将得到妥善积极的治疗。
- (4) 我参加本研究完全是自愿的,我可以拒绝参加或在任何时间退出研究,而不会遭到歧视 或报复,我的医疗待遇与权益亦不会受影响。

# 同时我声明:

- (1) 我愿意遵守研究流程;
- (2) 在研究期间,我愿意配合医生在规定的时间内就诊,并做相应的检查;
- (3) 已收到此份知情同意书。

研究参与者签字: 联系方式:

签字日期: 年 月 日 时 分

如果研究参与者为无/限制民事行为能力人(18岁以下的未成年人、丧失意识或各种原因导致思维障碍无法签署知情同意书时),请其监护人在此签名:

监护人签字: 与研究参与者的关系: 联系方式:

签字日期: 年 月 日 时 分

如果研究参与者/监护人无阅读能力,无法签署知情同意书时,请公正见证人在此签名:

公正见证人签字: 联系方式:

签字日期: 年 月 日 时 分

#### 研究者声明

我本人已向该研究参与者充分解释和说明了本研究的目的、研究方法、操作流程以及研

究参与者参加该研究可能存在的风险和潜在的利益,并满意地回答了研究参与者的所有有关 问题。

研究者(对研究参与者进行告知者)签名: 联系方式:

签字日期: 年 月 日 时 分